CLINICAL TRIAL: NCT05551390
Title: Effect of One-time Versus Three-times of Umbilical Cord Milking on Neonatal Hemoglobin in Late Preterm: A Randomized Controlled Trial
Brief Title: Effect of One-time Versus Three-times of Umbilical Cord Milking on Neonatal Hemoglobin in Late Preterm
Acronym: RRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 010/2564
Record Dates: First submitted 2022-09-06; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Umbilical Cord Milking

STUDY DESIGN:
Intervention Model Description: Late preterm pregnant women (34-36+6 week's gestation) that exclude placenta accrete/percreta, placenta previa, placental abruption, congenital anomaly and hydrops fetalis, were randomized in a 1:1 ratio to either one-time or three-times UCM.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- one-time umbilical cord milking (Experimental): Before UCM procedures, in the case of vaginal delivery, the maternity doctor or nurse held the newborn below the level of the introitus. In the case of a cesarean section, the surgeon carries the newborn below the level of the incision.
  Then maternity nurse or doctor swiped blood in length 20 centimeters of umbilical cord into the newborn, according to the number of swipes that assigned, then cutting the umbilical cord by the international standard methods. Newborns after birth were cared for and assessed according to the newborn nursing standards of QSMH in the department of pediatrics.
  Interventions: Other: one-time umbilical cord milking
- three-time umbilical cord milking (Experimental): Before UCM procedures, in the case of vaginal delivery, the maternity doctor or nurse held the newborn below the level of the introitus. In the case of a cesarean section, the surgeon carries the newborn below the level of the incision.
  Then maternity nurse or doctor swiped blood in length 20 centimeters of umbilical cord into the newborn, according to the number of swipes that assigned, then cutting the umbilical cord by the international standard methods. Newborns after birth were cared for and assessed according to the newborn nursing standards of QSMH in the department of pediatrics.
  Interventions: Other: three-times umbilical cord milking

INTERVENTIONS:
Other: one-time umbilical cord milking — Before UCM procedures, in the case of vaginal delivery, the maternity doctor or nurse held the newborn below the level of the introitus. In the case of a cesarean section, the surgeon carries the newborn below the level of the incision.
  Then maternity nurse or doctor swiped blood in length 20 centimeters of umbilical cord into the newborn, according to the number of swipes that assigned, then cutting the umbilical cord by the international standard methods. Newborns after birth were cared for and assessed according to the newborn nursing standards of QSMH in the department of pediatrics.
  Arms: one-time umbilical cord milking
Other: three-times umbilical cord milking — Before UCM procedures, in the case of vaginal delivery, the maternity doctor or nurse held the newborn below the level of the introitus. In the case of a cesarean section, the surgeon carries the newborn below the level of the incision.
  Then maternity nurse or doctor swiped blood in length 20 centimeters of umbilical cord into the newborn, according to the number of swipes that assigned, then cutting the umbilical cord by the international standard methods. Newborns after birth were cared for and assessed according to the newborn nursing standards of QSMH in the department of pediatrics.
  Arms: three-time umbilical cord milking

SUMMARY:
To compare the neonatal hemoglobin (Hb) in late preterm between one-time versus three-times of umbilical cord milking (UCM)

DETAILED DESCRIPTION:
This was a double-blind randomized controlled trial that performed between May 2021 to March 2022 at the Obstetrics and Gynecology Department of Queen Savang Vadhana Memorial Hospital. Late preterm pregnant women (34-36+6 week's gestation) that exclude placenta accrete/percreta, placenta previa, placental abruption, congenital anomaly and hydrops fetalis, were randomized in a 1:1 ratio to either one-time or three-times UCM. The primary outcome was neonatal Hb level at 48-72 hour after birth.

ELIGIBILITY:
Inclusion Criteria:

* Late preterm pregnant women (34-36+6 week's gestation)

Exclusion Criteria:

* placenta accrete
* placenta percreta
* placenta previa
* placental abruption
* congenital anomaly
* hydrops fetalis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome was neonatal Hb level | 48-72 hour after birth
  neonatal Hb level

CONTACTS AND LOCATIONS:
Locations (1):
- Wachira Prachakittikul, Chon Buri, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: No